CLINICAL TRIAL: NCT00844194
Title: A 12 Weeks Open Label Two Parallel Groups Study to Assess the Efficacy of Orally Administered Duloxetine 60 mg and 120 mg Per Day on Treatment Outcomes in Patients With Diabetic Peripheral Neuropathic Pain With and Without Co-morbid Major Depressive Disorder. The Primary Objective of This Study is to Evaluate Whether the Efficacy of Duloxetine Given as 60 mg to 120 mg Once Daily (QD), Measured by the BPI Interference Score After 12 Weeks Shows a Clinically Relevant Improvement in the DPNP Patients With Co-morbid MDD
Brief Title: Duloxetine in Patients With Diabetic in Peripheral Neuropathic Pain With or Without Co-morbid Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1208.34; 2008-002731-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Neuropathies; Depressive Disorder, Major
MeSH Terms: conditions — Diabetic Neuropathies; Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

ARMS (4):
- DPNP with depression (1) (Other): Patients that have diabetic polyneuropathy and depression and are responder to 60 mg duloxetine QD (>30% pain reduction after week 6)
  Interventions: Drug: Duloxetine 60 mg QD; Drug: Duloxetine 30 mg QD
- DPNP with depression (2) (Other): Patients that have diabetic polyneuropathy and depression and are non-responder to 60 mg duloxetine QD (<30% pain reduction after week 6)
  Interventions: Drug: Duloxetine 90 mg QD; Drug: Duloxetine 60 mg QD; Drug: Duloxetine 30 mg QD; Drug: Duloxetine 120 mg QD
- DPNP without depression (1) (Other): Patients that have diabetic polyneuropathy and no depression and are responder to 60 mg duloxetine QD (>30% pain reduction after week 6)
  Interventions: Drug: Duloxetine 60 mg QD; Drug: Duloxetine 30 mg QD
- DPNP without depression (2) (Other): Patients that have diabetic polyneuropathy and no depression and are non-responder to 60 mg duloxetine QD (<30% pain reduction after week 6)
  Interventions: Drug: Duloxetine 90 mg QD; Drug: Duloxetine 60 mg QD; Drug: Duloxetine 120 mg QD; Drug: Duloxetine 30 mg QD

INTERVENTIONS:
Drug: Duloxetine 60 mg QD — given to (1) all patients week 2-6; (2) all responders of both arms week 7-12
  Arms: DPNP without depression (1)
Drug: Duloxetine 60 mg QD — given to (1) all patients week 2-6; (2) all responders of both arms week 7-12
  Arms: DPNP with depression (1)
Drug: Duloxetine 30 mg QD — given to (1) all patients for one week as taper in; (2) all patients for taper down (responder for 2 weeks)
  Arms: DPNP without depression (1)
Drug: Duloxetine 30 mg QD — given to (1) all patients for one week as taper in; (2) all patients for taper down (responder for 2 weeks)
  Arms: DPNP with depression (1)
Drug: Duloxetine 90 mg QD — given to non-responders of both arms from day of notice that 120 mg is not tolerated to week 12 as 60 mg+30 mg Duloxetine QD
  Arms: DPNP with depression (2)
Drug: Duloxetine 90 mg QD — given to non-responders of both arms from day of notice that 120 mg is not tolerated to week 12 as 60 mg+30 mg Duloxetine QD
  Arms: DPNP without depression (2)
Drug: Duloxetine 60 mg QD — given to (1) all patients week 2-6; (2) all non-responders of both arms for first week of taper down
  Arms: DPNP without depression (2)
Drug: Duloxetine 60 mg QD — given to (1) all patients week 2-6; (2) all non-responders of both arms for first week of taper down
  Arms: DPNP with depression (2)
Drug: Duloxetine 120 mg QD — given to non-responders of both arms from week 7-12 as 2x60 mg Duloxetine QD, if tolerated
  Arms: DPNP without depression (2)
Drug: Duloxetine 30 mg QD — given to (1) all patients for one week as taper in; (2) all patients for taper down (non-responder for the second week of taper down)
  Arms: DPNP without depression (2)
Drug: Duloxetine 30 mg QD — given to (1) all patients for one week as taper in; (2) all patients for taper down (non-responder for the second week of taper down)
  Arms: DPNP with depression (2)
Drug: Duloxetine 120 mg QD — given to non-responders of both arms from week 7-12 as 2x60 mg Duloxetine QD, if tolerated
  Arms: DPNP with depression (2)

SUMMARY:
The primary objective is to evaluate, separately in diabetic polyneuropathic pain (DPNP) patients with and without co-morbid major depressive disorder (MDD), whether duloxetine given as 60 mg to 120 mg once daily (QD) leads to a clinically relevant improvement as measured by the change in Brief Pain Inventory (BPI) 24 hours average interference score from baseline to after 12 weeks. A clinically relevant improvement will be demonstrated if the confidence interval for the mean change from baseline does not lie above the clinically relevant change of -1.35. If statistically significant results are obtained for the DPNP patients with MDD, then the same evaluation will be performed for the DPNP patients without MDD in another confirmatory analysis.

As secondary objectives the study will compare the two groups (MDD+/MDD-) regarding efficacy of duloxetine on BPI severity scales, the distribution of different percentages of pain reduction among the patient population, and the patients and physicians impressions of severity and improvement of pain.

The study will also compare treatment outcomes regarding patient-relevant functionality and quality of life (QoL) between the two groups (MDD+/MDD-) by evaluating each single BPI interference item, the Short Form 12 (SF-12) Health Questionnaire and the West Haven Multidimensional Pain Inventory (MPI).

As a third group of secondary objectives the efficacy of duloxetine of the psychological symptoms (e.g. depression) of DPNP patients with or without depression will be assessed using the Hamilton depression scale, the Beck Depression Inventory-II and the hospital Anxiety and Depression Scale.

Further the effect of duloxetine treatment on fasting blood glucose (FBG) and hemoglobin A1c (HbA1c) will be evaluated.

To monitor safety and tolerability, treatment discontinuation rates, treatment emergent adverse events, change in vital signs, laboratory results and suicidal thoughts will be assessed.

ELIGIBILITY:
Inclusion criteria:

1. Present with pain due to bilateral peripheral neuropathy (according to International Statistical Classification of Diseases and Related Health Problems 10 (ICD 10).
2. To qualify for the MDD+ cohort, patients need to meet the ICD-10 criteria for MDD. Furthermore, Hamilton rating scale for depression 17 (HAMD-17) scores need to match with the ICD-10 criteria for qualification of the MDD+ or MDD- groups.
3. Male or female outpatients at least 18 years of age.
4. Females with child bearing potential must test negative for a serum pregnancy test at Visit 1. Females of child-bearing potential (not surgically sterilized and between menarche and 1 year post-menopause) must agree to utilize medically acceptable and reliable means of birth control as determined by the investigator during the study and for 1 month following the last dose of the study. Examples of reliable methods include use of oral contraceptives or Depo-Clinovir Contraceptive Injection (sterile medroxyprogesterone acetate suspension, Pharmacia), partner with vasectomy, diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms with contraceptive foam, or intrauterine devices. Women who are pregnant or breast-feeding may not participate in the study.
5. Educational level and degree of understanding such that they can communicate intelligibly with the investigator and study coordinator.
6. Judged to be reliable and agrees to keep all appointments for clinic visits, tests, and procedures required by the protocol.

Exclusion criteria:

1. Have already a diagnosis of Depression and are currently treated with an antidepressant medication for depression, when entering the study.
2. Suffer from pain that cannot be clearly differentiated from or conditions that interfere with the assessment of DPNPain.
3. Had a historical exposure to drugs known to cause neuropathy, that could have been responsible for neuropathy.
4. Have previously been treated with duloxetine (for DPNP or MDD)
5. Are judged to be at suicidal risk by the clinical investigator or as defined by a score of 2 or greater on question 9 of the Beck Depression Inventory-II (BDI-II).
6. Had a history of substance abuse or dependence within the past year, excluding nicotine and caffeine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (25):
- Germany (25):
  - 1208.34.49008 Boehringer Ingelheim Investigational Site, Achim Bei Bremen
  - 1208.34.49025 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1208.34.49001 Boehringer Ingelheim Investigational Site, Bad Mergentheim
  - 1208.34.49018 Boehringer Ingelheim Investigational Site, Baesweiler
  - 1208.34.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1208.34.49005 Boehringer Ingelheim Investigational Site, Berlin
  - 1208.34.49009 Boehringer Ingelheim Investigational Site, Berlin
  - 1208.34.49021 Boehringer Ingelheim Investigational Site, Bremen
  - 1208.34.49028 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1208.34.49012 Boehringer Ingelheim Investigational Site, Gera
  - 1208.34.49004 Boehringer Ingelheim Investigational Site, Hamburg
  - 1208.34.49020 Boehringer Ingelheim Investigational Site, Hamburg
  - 1208.34.49023 Boehringer Ingelheim Investigational Site, Hamburg
  - 1208.34.49015 Boehringer Ingelheim Investigational Site, Hattingen
  - 1208.34.49027 Boehringer Ingelheim Investigational Site, Heidenheim
  - 1208.34.49016 Boehringer Ingelheim Investigational Site, Kelkheim
  - 1208.34.49006 Boehringer Ingelheim Investigational Site, Limburgerhof
  - 1208.34.49022 Boehringer Ingelheim Investigational Site, Münster
  - 1208.34.49019 Boehringer Ingelheim Investigational Site, Neuwied
  - 1208.34.49024 Boehringer Ingelheim Investigational Site, Saint Ingberg
  - 1208.34.49007 Boehringer Ingelheim Investigational Site, Steglitz
  - 1208.34.49010 Boehringer Ingelheim Investigational Site, Stuhr
  - 1208.34.49013 Boehringer Ingelheim Investigational Site, Unterhaching
  - 1208.34.49029 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 1208.34.49026 Boehringer Ingelheim Investigational Site, Wuppertal

RESULTS

PARTICIPANT FLOW:
Groups:
- Without Major Depressive Disorder (MDD-): Patients with diabetic polyneuropathy and no depression
- With Major Depressive Disorder (MDD+): Patients with diabetic polyneuropathy and depression
Period: Overall Study
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Started | 78 | 30
Completed | 53 | 22
Not Completed | 25 | 8
Not completed — Adverse Event | 17 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 3 | 0
Not completed — Other reason (not specified) | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients receiving at least one dose of study medication (TS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+) | Total
Number analyzed (Participants) | 78 | 30 | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (10.2) | 66.6 (9.8) | 67.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 15 | 51
  Male | 42 | 15 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change of Brief Pain Inventory (BPI) Average Interference Score From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The BPI average interference score ranges from 0 (pain does not interfere) to 10 (pain completely interferes).
Time Frame: Baseline and Week 12
Population: All patients receiving at least one dose of study medication, having any efficacy data and dosage of duloxetine was not more than 60mg before visit 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -1.4 (1.91) | -2.2 (2.2)
Statistical Analysis 1: Comparison: Without Major Depressive Disorder (MDD-); Test type: Superiority or Other; p < 0.0001, ANCOVA; with last observation carried forward (LOCF); LSmean = -1.49, 95% CI 2-sided [-1.89 to -1.10]
Statistical Analysis 2: Comparison: With Major Depressive Disorder (MDD+); Test type: Superiority or Other; p < 0.0001, ANCOVA; LSmean = -1.67, 95% CI 2-sided [-2.30 to -1.04]

2. Secondary Outcome: Change of Brief Pain Inventory (BPI) Average Interference Score From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The BPI average interference score ranges from 0 (pain does not interfere) to 10 (pain completely interferes).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -1.2 (1.88) | -2.0 (1.96)

3. Secondary Outcome: Change in BPI Worst Pain During Treatment From Baseline to Week 2
Description: The change from baseline reflects the week 2 value minus the baseline value. The BPI pain ranges from 0 (no pain) to 10 (pain as bad as the patient can imagine).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -2.2 (2.27) | -1.9 (2.19)

4. Secondary Outcome: Change in Worst Pain (BPI) From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The BPI pain ranges from 0 (no pain) to 10 (pain as bad as the patient can imagine).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -2.6 (2.36) | -3.3 (2.56)

5. Secondary Outcome: Change in Worst Pain (BPI) From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The BPI pain ranges from 0 (no pain) to 10 (pain as bad as the patient can imagine).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 64 | 26
Scores on a scale | -2.8 (2.55) | -3.2 (3.41)

6. Secondary Outcome: Change in Least Pain (BPI) From Baseline to Week 2
Description: as for outcome 3
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -1.1 (2.35) | -0.2 (1.7)

7. Secondary Outcome: Change in Least Pain During Treatment (BPI) From Baseline to Week 6
Description: as for outcome 4
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -1.7 (1.92) | -1.3 (2.1)

8. Secondary Outcome: Change in Least Pain (BPI) From Baseline to Week 12
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -1.5 (2.13) | -1.1 (2.07)

9. Secondary Outcome: Change in Average Pain (BPI) From Baseline to Week 2
Description: as for outcome 3
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -1.6 (1.87) | -1.1 (1.63)

10. Secondary Outcome: Change in Average Pain During Treatment (BPI) From Baseline to Week 6
Description: as for outcome 4
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -2.6 (1.92) | -2.6 (2.0)

11. Secondary Outcome: Change in Average Pain (BPI) From Baseline to Week 12
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -2.4 (1.88) | -2.2 (2.07)

12. Secondary Outcome: Number of Patients With a Reduction in BPI Average Pain at Week 2
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 71 | 30
Participants
  >=30% | 29 | 9
  >=50% | 19 | 3
  Missing | 5 | 2

13. Secondary Outcome: Number of Patients With a Reduction in BPI Average Pain at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 71 | 30
Participants
  >=30% | 42 | 17
  >=50% | 30 | 12
  Missing | 14 | 6

14. Secondary Outcome: Number of Patients With a Reduction in BPI Average Pain at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 71 | 30
Participants
  >=30% | 42 | 17
  >=50% | 30 | 11
  Missing | 6 | 4

15. Secondary Outcome: Change in Pain During Treatment (BPI) From Baseline to Week 2
Description: The change from baseline reflects the pain at week 2 minus the pain at baseline. The BPI pain ranges from 0 (no pain) to 10 (pain as bad as the patient can imagine).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -1.4 (2.34) | -1.0 (2.06)

16. Secondary Outcome: Change in Pain (BPI) From Baseline to Week 6
Description: The change from baseline reflects the pain at week 6 minus the pain at baseline. The BPI pain ranges from 0 (no pain) to 10 (pain as bad as the patient can imagine).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -2.0 (2.27) | -1.7 (3.01)

17. Secondary Outcome: Change in Pain During Treatment (BPI) From Baseline to Week 12
Description: The change from baseline reflects the pain at week 12 minus the pain at baseline. The BPI pain ranges from 0 (no pain) to 10 (pain as bad as the patient can imagine).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -1.7 (2.6) | -1.5 (2.21)

18. Secondary Outcome: Change in Relief of Pain (BPI) From the Week Before Baseline to the Week Before Week 2
Description: The change from baseline reflects the week 2 value minus the baseline value. The relief of pain ranges from 0% (no relief) to 100% (complete relief).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 62 | 25
scores on a scale | 21.5 (33.87) | 18.0 (35.0)

19. Secondary Outcome: Change in Relief of Pain (BPI) From the Week Before Baseline to the Week Before Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The relief of pain ranges from 0% (no relief) to 100% (complete relief).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 51 | 23
scores on a scale | 23.5 (37.3) | 31.7 (45.49)

20. Secondary Outcome: Change in Relief of Pain (BPI) From the Week Before Baseline to the Week Before Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The relief of pain ranges from 0% (no relief) to 100% (complete relief).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 54 | 24
scores on a scale | 30.2 (35.85) | 22.9 (33.55)

21. Secondary Outcome: Change in Interference of Pain With General Activity (BPI) From Baseline to Week 2
Description: The change from baseline reflects the week 2 value minus the baseline value. The BPI interference score ranges from 0 (pain does not interfere) to 10 (pain completely interferes).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 67 | 28
Scores on a scale | -1.6 (2.5) | -1.1 (2.02)

22. Secondary Outcome: Change in Interference of Pain With General Activity (BPI) From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The BPI interference score ranges from 0 (pain does not interfere) to 10 (pain completely interferes).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -1.8 (2.89) | -2.5 (3.16)

23. Secondary Outcome: Change in Interference of Pain With General Activity (BPI) From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The BPI interference score ranges from 0 (pain does not interfere) to 10 (pain completely interferes).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -2.4 (2.53) | -2.7 (2.76)

24. Secondary Outcome: Change in Interference of Pain With Mood (BPI) From Baseline to Week 2
Description: as for outcome 21
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -1.1 (2.3) | -1.5 (1.73)

25. Secondary Outcome: Change in Interference of Pain With Mood (BPI) From Baseline to Week 6
Description: as for outcome 22
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -1.4 (2.4) | -3.1 (3.08)

26. Secondary Outcome: Change in Interference of Pain With Mood (BPI) From Baseline to Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -1.2 (2.68) | -3.0 (3.28)

27. Secondary Outcome: Change in Interference of Pain With Walking Ability (BPI) From Baseline to Week 2
Description: as for outcome 21
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -0.9 (2.03) | -1.0 (2.19)

28. Secondary Outcome: Change in Interference of Pain With Walking Ability (BPI) From Baseline to Week 6
Description: as for outcome 22
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 56 | 24
Scores on a scale | -1.3 (2.55) | -2.1 (3.26)

29. Secondary Outcome: Change in Interference of Pain With Walking Ability (BPI) From Baseline to Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -1.9 (2.86) | -2.4 (3.11)

30. Secondary Outcome: Change in Interference of Pain With Normal Work (BPI) From Baseline to Week 2
Description: as for outcome 21
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 28
Scores on a scale | -0.9 (1.76) | -0.1 (2.34)

31. Secondary Outcome: Change in Interference of Pain With Normal Work (BPI) From Baseline to Week 6
Description: as for outcome 22
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -1.1 (2.47) | -1.3 (2.92)

32. Secondary Outcome: Change in Interference of Pain With Normal Work (BPI) From Baseline to Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 64 | 26
Scores on a scale | -1.4 (1.89) | -1.8 (2.67)

33. Secondary Outcome: Change in Interference of Pain With Relations to Other People (BPI) From Baseline to Week 2
Description: as for outcome 21
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 67 | 28
Scores on a scale | -0.5 (2.68) | -0.1 (2.80)

34. Secondary Outcome: Change in Interference of Pain With Relations to Other People (BPI) From Baseline to Week 6
Description: as for outcome 22
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -0.6 (2.64) | -1.7 (2.60)

35. Secondary Outcome: Change in Interference of Pain With Relations to Other People (BPI) From Baseline to Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 64 | 26
Scores on a scale | -0.4 (2.42) | -1.7 (2.71)

36. Secondary Outcome: Change in Interference of Pain With Sleep (BPI) From Baseline to Week 2
Description: as for outcome 21
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -0.8 (3.21) | -1.0 (2.46)

37. Secondary Outcome: Change in Interference of Pain With Sleep (BPI) From Baseline to Week 6
Description: as for outcome 22
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -1.1 (3.50) | -1.5 (3.44)

38. Secondary Outcome: Change in Interference of Pain With Sleep (BPI) From Baseline to Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -1.5 (2.53) | -1.9 (3.05)

39. Secondary Outcome: Change in Interference of Pain With Enjoyment of Life (BPI) From Baseline to Week 2
Description: as for outcome 21
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 67 | 28
Scores on a scale | -0.7 (2.06) | -0.6 (1.97)

40. Secondary Outcome: Change in Interference of Pain With Enjoyment of Life (BPI) From Baseline to Week 6
Description: as for outcome 22
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -1.2 (2.52) | -2.2 (2.90)

41. Secondary Outcome: Change in Interference of Pain With Enjoyment of Life (BPI) From Baseline to Week 12
Description: as for outcome 23
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -0.9 (2.93) | -2.1 (2.30)

42. Secondary Outcome: Patient Global Impression - Improvement (PGI-I) at Week 2
Description: The investigator judged the improvement of the patient's global impression during treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 67 | 28
Scores on a scale | 3.0 (1.01) | 3.2 (0.82)

43. Secondary Outcome: Patient Global Impression - Improvement (PGI-I) at Week 6
Description: as for outcome 42
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 23
Scores on a scale | 2.5 (0.87) | 2.5 (1.04)

44. Secondary Outcome: Patient Global Impression - Improvement (PGI-I) at Week 12
Description: as for outcome 42
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 64 | 26
Scores on a scale | 2.5 (1.35) | 2.7 (1.29)

45. Secondary Outcome: Change in Beck Depression Inventory Total Score (BDI-II) From Baseline to Week 2
Description: The change from baseline reflects the week 2 value minus the baseline value. The BDI-II total score ranges from 0 to 63, with a higher score indicating a higher level of depression.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 63 | 26
Scores on a scale | -0.9 (3.61) | -3.1 (5.79)

46. Secondary Outcome: Change in Beck Depression Inventory Total Score (BDI-II) From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The BDI-II total score ranges from 0 to 63, with a higher score indicating a higher level of depression.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 50 | 23
Scores on a scale | -1.8 (5.93) | -7.3 (7.05)

47. Secondary Outcome: Change in Beck Depression Inventory Total Score (BDI-II) From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The BDI-II total score ranges from 0 to 63, with a higher score indicating a higher level of depression.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 58 | 24
Scores on a scale | -1.6 (6.02) | -7.8 (7.25)

48. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) Anxiety Total Score From Baseline to Week 2
Description: The change from baseline reflects the week 2 value minus the baseline value. The HADS anxiety total score ranges from 0 (no anxiety) to 21 (extreme anxiety).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 67 | 28
Scores on a scale | -0.7 (2.23) | -1.2 (2.94)

49. Secondary Outcome: Change in HADS Anxiety Total Score From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The HADS anxiety total score ranges from 0 (no anxiety) to 21 (extreme anxiety).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 56 | 24
Scores on a scale | -0.8 (2.98) | -2.2 (3.03)

50. Secondary Outcome: Change in HADS Anxiety Total Score From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The HADS anxiety total score ranges from 0 (no anxiety) to 21 (extreme anxiety).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -1.0 (3.03) | -3.3 (4.08)

51. Secondary Outcome: Change in HADS Depression Total Score From Baseline to Week 2
Description: The change from baseline reflects the week 2 value minus the baseline value. The HADS depression total score ranges from 0 (no depression) to 21 (extreme depression).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -0.5 (1.65) | -1.6 (3.21)

52. Secondary Outcome: Change in HADS Depression Total Score From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The HADS depression total score ranges from 0 (no depression) to 21 (extreme depression).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 55 | 24
Scores on a scale | -0.8 (2.80) | -3.4 (3.78)

53. Secondary Outcome: Change in HADS Depression Total Score From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The HADS depression total score ranges from 0 (no depression) to 21 (extreme depression).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 64 | 26
Scores on a scale | -0.7 (3.07) | -3.7 (3.92)

54. Secondary Outcome: Change in Short Form Health Survey (SF-12) - Physical Component Summary From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. A lower score corresponds to a lower level of physical health. Values can range from 0 to 100.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 45 | 18
Scores on a scale | 4.0 (8.37) | -0.0 (11.74)

55. Secondary Outcome: Change in Short Form Health Survey (SF-12) - Physical Component Summary From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. A lower score corresponds to a lower level of physical health. Values can range from 0 to 100.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 49 | 21
Scores on a scale | 3.5 (9.64) | 2.4 (11.51)

56. Secondary Outcome: Change in Short Form Health Survey (SF-12) - Mental Component Summary From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. A lower score corresponds to a lower level of mental health. Values can range from 0 to 100.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 45 | 18
Scores on a scale | -0.9 (8.19) | 5.0 (11.11)

57. Secondary Outcome: Change in Short Form Health Survey (SF-12) - Mental Component Summary From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. A lower score corresponds to a lower level of mental health. Values can range from 0 to 100.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 49 | 21
Scores on a scale | 0.7 (10.19) | 6.0 (13.07)

58. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Interference of Pain (With Subjective Well-being) From Baseline to Week 6
Description: Pain-related life interference (with family and marital functioning, work, social activities). The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (no interference) to 6 (extreme interference).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 56 | 24
Scores on a scale | -1.0 (1.06) | -0.9 (1.24)

59. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Interference of Pain From Baseline to Week 12
Description: Pain-related life interference (with family and marital functioning, work, social activities). The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (no interference) to 6 (extreme interference).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 64 | 26
Scores on a scale | -1.1 (1.13) | -1.0 (1.37)

60. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Support From Baseline to Week 6
Description: Appraisal of support received from spouse, family and significant others. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (no support) to 6 (very much support).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 54 | 22
Scores on a scale | -0.4 (1.28) | 0.5 (1.59)

61. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Support Which the Patient Received From Baseline to Week 12
Description: Appraisal of support received from spouse, family and significant others. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (no support) to 6 (very much support).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 59 | 24
Scores on a scale | -0.2 (1.54) | 0.4 (1.90)

62. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Pain Severity From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (not at all strong) to 6 (very strong).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 55 | 24
Scores on a scale | -1.2 (1.34) | -1.0 (1.33)

63. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Pain Severity From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (no control) to 6 (extreme control).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 61 | 26
Scores on a scale | -1.5 (1.39) | -1.2 (1.35)

64. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Life Control From Baseline to Week 6
Description: Perceived life control and ability to solve problems and feelings of personal mastery and competence. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (no control) to 6 (extreme control).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 55 | 24
Scores on a scale | 0.2 (1.14) | 0.2 (1.16)

65. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Life Control From Baseline to Week 12
Description: Perceived life control and ability to solve problems and feelings of personal mastery and competence. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (no control) to 6 (extreme control).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 62 | 25
Scores on a scale | 0.4 (1.10) | 0.3 (1.57)

66. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Affective Distress From Baseline to Week 6
Description: Affective distress, including ratings of depressed mood, irritability, and tension. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (no distress) to 6 (extreme distress).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 56 | 24
Scores on a scale | -0.3 (1.01) | -0.5 (1.04)

67. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Affective Distress From Baseline to Week 12
Description: Affective distress, including ratings of depressed mood, irritability, and tension. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (no distress) to 6 (extreme distress).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 62 | 26
Scores on a scale | -0.5 (1.00) | -0.8 (1.13)

68. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Negative Responses From Baseline to Week 6
Description: Degree to which significant others display negative responses to the patient's pain behaviors and complaints. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 54 | 24
Scores on a scale | -0.1 (0.87) | -0.7 (2.16)

69. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Negative Responses From Baseline to Week 12
Description: Degree to which significant others display negative responses to the patient's pain behaviors and complaints. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 62 | 26
Scores on a scale | 0.1 (0.73) | -0.3 (2.03)

70. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Solicitous Responses From Baseline to Week 6
Description: Degree to which significant others display solicitous responses to the patient's pain behaviors and complaints. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 54 | 24
Scores on a scale | -0.2 (1.12) | -0.2 (2.08)

71. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Solicitous Responses From Baseline to Week 12
Description: Degree to which significant others display solicitous responses to the patient's pain behaviors and complaints. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 62 | 26
Scores on a scale | -0.2 (1.10) | 0.2 (2.30)

72. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Degree to Which Significant Others Display Distracting Responses to the Patient's Pain Behaviors and Complaints From Baseline to Week 6
Description: Degree to which significant others display distracting responses to the patient's pain behaviors and complaints. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 53 | 24
Scores on a scale | -0.1 (1.35) | -0.1 (2.25)

73. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Degree to Which Significant Others Display Distracting Responses to the Patient's Pain Behaviors and Complaints From Baseline to Week 12
Description: Degree to which significant others display distracting responses to the patient's pain behaviors and complaints. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 62 | 26
Scores on a scale | -0.2 (1.19) | 0.0 (2.43)

74. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Household Chores From Baseline to Week 6
Description: Frequency with which the patient engages in household chores. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | 0.0 (1.24) | -0.1 (0.79)

75. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Household Chores From Baseline to Week 12
Description: Frequency with which the patient engages in household chores. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | 0.1 (1.29) | -0.1 (0.99)

76. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Outdoor Work From Baseline to Week 6
Description: Frequency with which the patient engages in outdoor work. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 54 | 21
Scores on a scale | -1.2 (6.29) | 0.3 (2.01)

77. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Outdoor Work From Baseline to Week 12
Description: Frequency with which the patient engages in outdoor work. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 62 | 24
Scores on a scale | -1.6 (10.24) | 0.6 (2.37)

78. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Social Activities From Baseline to Week 6
Description: Frequency with which the patient engages in social activities. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | 0.1 (0.80) | 0.1 (0.70)

79. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): Social Activities From Baseline to Week 12
Description: Frequency with which the patient engages in social activities. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | 0.1 (0.64) | 0.3 (1.11)

80. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): General Activities From Baseline to Week 6
Description: Frequency with which the patient engages in general activities. The change from baseline reflects the week 6 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -0.2 (1.66) | 0.1 (0.60)

81. Secondary Outcome: Change in Multidimensional Pain Inventory (MPI): General Activities From Baseline to Week 12
Description: Frequency with which the patient engages in general activities. The change from baseline reflects the week 12 value minus the baseline value. The scores range from 0 (never) to 6 (very frequently).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Scores on a scale | -0.3 (2.73) | 0.3 (0.95)

82. Secondary Outcome: Change in Clinical Global Impression - Severity Pain From Baseline to Week 2
Description: The change from baseline reflects the week 2 value minus the baseline value. The score of the Clinical global impression ranges from 1 (not ill at all) to 7 (extremely ill).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 28
Scores on a scale | -0.5 (0.96) | -0.4 (0.62)

83. Secondary Outcome: Change in Clinical Global Impression - Severity Pain From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. The score of the Clinical global impression ranges from 1 (not ill at all) to 7 (extremely ill).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores on a scale | -0.7 (1.02) | -0.8 (0.78)

84. Secondary Outcome: Change in Clinical Global Impression - Severity Pain From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. The score of the Clinical global impression ranges from 1 (not ill at all) to 7 (extremely ill).
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: Scores of a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 27
Scores of a scale | -0.8 (1.08) | -1.0 (0.94)

85. Secondary Outcome: Change in Hamilton Depression Score From Baseline to Week 2
Description: The change from baseline reflects the week 2 value minus the baseline value. A lower score corresponds to a lower level of depression. The score ranges from 0 to 52.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 28
Scores on a scale | -0.2 (2.50) | -4.5 (5.29)

86. Secondary Outcome: Change in Hamilton Depression Score From Baseline to Week 6
Description: The change from baseline reflects the week 6 value minus the baseline value. A lower score corresponds to a lower level of depression. The score ranges from 0 to 52.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores of a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 57 | 24
Scores of a scale | -1.5 (2.89) | -9.3 (4.99)

87. Secondary Outcome: Change in Hamilton Depression Score From Baseline to Week 12
Description: The change from baseline reflects the week 12 value minus the baseline value. A lower score corresponds to a lower level of depression. The score ranges from 0 to 52.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 27
Scores on a scale | -0.8 (3.30) | -9.7 (5.50)

88. Secondary Outcome: Suicidal Thoughts by BDI-II at Week 2
Time Frame: Week 2
Population: All patients receiving at least one dose of study medication and having data at week 2.
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 70 | 28
Participants
  No thoughts of killing myself | 67 | 27
  Thoughts of killing myself | 3 | 1
  Like to kill myself | 0 | 0
  Kill myself if chance | 0 | 0
  Missing | 0 | 0

89. Secondary Outcome: Suicidal Thoughts by BDI-II at Week 6
Time Frame: Week 6
Population: All patients receiving at least one dose of study medication and having data at week 6.
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 59 | 24
Participants
  No thoughts of killing myself | 57 | 22
  Thoughts of killing myself | 2 | 1
  Like to kill myself | 0 | 0
  Kill myself if chance | 0 | 0
  Missing | 0 | 1

90. Secondary Outcome: Suicidal Thoughts by BDI-II at Week 12
Time Frame: Week 12
Population: All patients receiving at least one dose of study medication and having data at week 12.
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 65 | 26
Participants
  No thoughts of killing myself | 63 | 24
  Thoughts of killing myself | 0 | 2
  Like to kill myself | 0 | 0
  Kill myself if chance | 0 | 0
  Missing | 2 | 0

91. Secondary Outcome: Suicidal Thoughts or Behaviours by HAMD-17 at Week 2
Time Frame: Week 2
Population: All patients receiving at least one dose of study medication and having data at week 2.
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 68 | 28
Participants
  Absent | 68 | 26
  Feels life is not worth living | 0 | 2
  Thoughts of possible death to self | 0 | 0
  Suicidal ideas or gestures | 0 | 0
  Attempts at suicide | 0 | 0
  Missing | 0 | 0

92. Secondary Outcome: Suicidal Thoughts or Behaviours by HAMD-17 at Week 6
Time Frame: Week 6
Population: All patients receiving at least one dose of study medication and having data at week 6.
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 60 | 24
Participants
  Absent | 60 | 22
  Feels life is not worth living | 0 | 2
  Thoughts of possible death to self | 0 | 0
  Suicidal ideas or gestures | 0 | 0
  Attempts at suicide | 0 | 0
  Missing | 0 | 0

93. Secondary Outcome: Suicidal Thoughts or Behaviours by HAMD-17 at Week 12
Time Frame: Week 12
Population: All patients receiving at least one dose of study medication and having data at week 12.
Measure: Number; unit: Participants
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 27
Participants
  Absent | 66 | 26
  Feels life is not worth living | 0 | 1
  Thoughts of possible death to self | 0 | 0
  Suicidal ideas or gestures | 0 | 0
  Attempts at suicide | 0 | 0
  Missing | 0 | 0

94. Secondary Outcome: Change of Fasting Blood Glucose From Baseline at Week 12
Description: Ancova analysis controlling for baseline and insulin intake
Time Frame: Baseline and Week 12
Population: All patients receiving at least one dose of study medication and having data of fasting blood glucose at baseline and at week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 42 | 15
mg/dL | 14.9 [-12.0 to 41.8] | 13.0 [-37.7 to 63.7]

95. Secondary Outcome: Change of Glycosylated Hemoglobin A1c (HbA1c) From Baseline at Week 12
Description: Ancova analysis controlling for baseline and insulin intake
Time Frame: Baseline and Week 12
Population: All patients receiving at least one dose of study medication and having data of HbA1c at baseline and at week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 66 | 27
percent | 0.1 [-0.1 to 0.3] | 0.1 [-0.3 to 0.4]

96. Secondary Outcome: Change of Systolic Blood Pressure From Baseline at Week 12
Time Frame: Baseline and Week 12
Population: All patients receiving at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 75 | 30
mmHg | -0.4 (16.04) | -2.8 (17.40)

97. Secondary Outcome: Change of Diastolic Blood Pressure From Baseline at Week 12
Time Frame: Baseline and Week 12
Population: All patients receiving at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 75 | 30
mmHg | 2.2 (10.03) | -0.6 (8.86)

98. Secondary Outcome: Change of Pulse Rate From Baseline at Week 12
Time Frame: Baseline and Week 12
Population: All patients receiving at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Number analyzed (Participants) | 75 | 30
beats per minute (bpm) | 2.4 (9.53) | 2.9 (9.40)

99. Primary Outcome: Change of Brief Pain Inventory (BPI) Average Interference Score From Baseline to Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- MDD- Responder: MDD-, treatment responder. 60mg Duloxetine (DLX) for 12 weeks
- MDD+ Responder: MDD+, treatment responder. 60mg Duloxetine (DLX) for 12 weeks
- MDD- Non-Responder: MDD-, not treatment responder. 60mg, after week 5 120mg DLX
- MDD+ Non-Responder: MDD+, not treatment responder. 60mg, after week 5 120mg DLX
Arm/Group | MDD- Responder | MDD+ Responder | MDD- Non-Responder | MDD+ Non-Responder
Number analyzed (Participants) | 40 | 16 | 15 | 6
Scores on a scale | -1.7 (1.65) | -2.2 (2.0) | -0.9 (2.5) | -2.6 (3.31)

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: 12 Weeks treatment period (6 weeks for Treatment Phase 1 and 6 weeks for Treatment Phase 2) and a 2-week taper phase.
Arm/Group | Without Major Depressive Disorder (MDD-) | With Major Depressive Disorder (MDD+)
Serious Adverse Events (participants affected / at risk) | 4/78 | 2/30
Other Adverse Events (participants affected / at risk) | 28/78 | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Without Major Depressive Disorder (MDD-) (N=78) | With Major Depressive Disorder (MDD+) (N=30)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Without Major Depressive Disorder (MDD-) (N=78) | With Major Depressive Disorder (MDD+) (N=30)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 11 | 3
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 0
Fatigue (General disorders) | 4 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 2
Micturition disorder (Renal and urinary disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.